CLINICAL TRIAL: NCT00043862
Title: A Phase II Trial of Twice Daily Oral Topotecan as a Radiation Sensitizer With Twice Daily Radiotherapy for Newly Diagnosed Small Cell Lung Cancer
Brief Title: The Study Of An Oral Drug Called A Radiation Sensitizer In Patients With Newly Diagnosed Small Cell Lung Cancer (SCLC)
Acronym: (SCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104864/535
Record Dates: First submitted 2002-08-14; First posted 2002-08-15 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2013-03

CONDITIONS: Lung Cancer, Small Cell; Small Cell Lung Cancer
Keywords: Hycamtin; oral; Radiation Sensitization; Small Cell Lung Cancer; newly diagnosed; limited stage; topotecan
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: topotecan

SUMMARY:
This study will gather information on the effectiveness and safety of a treatment program for small cell lung cancer (SCLC) that uses an FDA approved chemotherapy combination, radiation therapy, and an oral investigational drug that may enhance the effects of radiation therapy. Study patients will receive two additional courses of the standard chemotherapy combination after completing radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have newly diagnosed, limited stage SCLC (small cell lung cancer), with no prior radiotherapy. Patients are allowed to have had a resection or biopsy.
* Women of reproductive potential must have a negative serum pregnancy test at the study screening visit.
* Patients must give written informed consent to participate in the study.
* Patients must be able to take oral medication.
* Patients should be completely recovered from recent surgery.
* Laboratory criteria: Patients must have adequate bone marrow reserve and adequate kidney and liver function.
* Patients must be evaluated by the radiation oncologist prior to study entry.

Exclusion Criteria:

* Extensive Stage SCLC.
* Women who are pregnant or lactating.
* Use of an investigational drug within 30 days prior to the first dose of study medication.
* Any medically/clinically significant active infection.
* Symptoms of the SCLC spreading to the brain.
* Patients with limited stage SCLC who have undergone complete resection with no measurable disease prior to starting chemotherapy.
* Severe medical problems, unrelated to SCLC, that would limit the patient's full ability to follow all study rules and procedures, or that would expose the patient to extreme risk.
* Other ongoing, immunotherapy or radiotherapy being administered at the time as study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2002-08; Primary Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Response rate

SECONDARY OUTCOMES:
Time to Progression, response duration, survival, quantitative and qualitative assessment of tolerability

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (30):
- United States (30):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Scarborough, Maine
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Duluth, Minnesota
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Robbinsdale, Minnesota
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Saint Louis, Montana
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Green Bay, Wisconsin
  - GSK Investigational Site, La Crosse, Wisconsin
  - GSK Investigational Site, Madison, Wisconsin
  - GSK Investigational Site, Milwaukee, Wisconsin
  - GSK Investigational Site, Wausau, Wisconsin